CLINICAL TRIAL: NCT05889728
Title: Assessment of the Diagnostic and Theranostic Potential of Ga Bombesin PET/CT (NeoB) Imaging for Staging of ER/PR + HER2- Breast Cancer Patients With Metastatic Disease: Comparison to Conventional Imaging
Brief Title: Pilot Trial to Assess 68Ga Bombesin PET/CT (NeoB) Imaging for Staging of Breast Cancer
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: St Vincent's Hospital, Sydney (Other)
Collaborators: Novartis (Industry)
Responsible Party: Principal Investigator, Louise Emmett, Professor, St Vincent's Hospital, Sydney
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: Best TRial
Record Dates: First submitted 2023-04-05; First posted 2023-06-05 (Actual); Last update posted 2023-06-05 (Actual); Status verified 2023-05

CONDITIONS: Breast Cancer
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Intervention Model Description: Female patients aged 18 or above with ER/PR+ HER2 - metastatic breast cancer presenting for standard of care staging/restaging prior to treatment of metastatic disease.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- 68Ga Bombesin PET/CT (NeoB) imaging for staging breast cancer (Experimental): All patients will undergo a single time point imaging at Day 0 with PET CT to be conducted 120 (+/- 30) minutes after intravenous administration with 68Ga NeoB (3.0MBq/kg or up to a maximum of 250 Mbq).
  Interventions: Drug: [68Ga]GA-NeoB

INTERVENTIONS:
Drug: [68Ga]GA-NeoB — Is a positron emission tomography (PET) imaging agent, intended as a selection tool for [177Lu]Lu-NeoB treatment in patients with tumors overexpressing gastrin releasing peptide receptor (GRPR).

SUMMARY:
This phase IIb pilot study will enrol 20 patients (women) presenting with metastatic breast cancer (ER/PR + HER2- on histology) who require imaging for staging or re-staging of their disease.

DETAILED DESCRIPTION:
There is little published literature evaluating the usefulness of Ga Bombesin-PET imaging in comparison to currently accepted imaging modalities for detecting progressive metastatic breast cancer. This study aims to produce preliminary research to evaluate its clinical value in breast cancer, given the promising previously published cell line and mouse work in ER/PR+ HER2- tumours. It further aims to ascertain the theranostic potential of the NeoB peptide in the ER/PR + Her 2- population, particularly assessing the level of heterogeneity at sites of active malignancy compared to FDG PET.

This study will add PET CT imaging using a tracer agent (NeoB) that directly targets the breast cancer cell. The ability of this new PET CT scan to detect sites of metastatic disease will be compared to standard procedures which include Diagnostic CT, bone scan and 18F-FDG PET.

All patients will undergo a single time point imaging at Day 0 with PET CT to be conducted 120 (+/- 30) minutes after intravenous administration with 68Ga NeoB (3.0MBq/kg).

ELIGIBILITY:
Inclusion Criteria:

* Female patients aged 18 or above
* Ability to provide informed consent documentation indicating that they understand the purpose of and procedures required for the study, and are willing to participate in the study
* Estrogen/Progesterone receptor +ve HER2 negative disease confirmed on prior biopsy (primary or metastatic site).
* Metastatic breast cancer being staged or re-staged prior to treatment of metastatic disease (including those presenting with up-front metastatic disease with primary breast cancer in-situ and those who have progressed on a line of treatment for metastatic breast cancer that are suitable for another line of treatment)
* Metastatic breast cancer being staged or restaged prior to change in treatment with standard imaging within 3 weeks of enrolment (CT CAP, bone scan, FDG PET CT)

Exclusion Criteria:

* Pregnancy or lactation (patients should use highly effective methods of contraception during and for 12h after administration)
* Significant inter-current acute illness as per investigator discretion that prevent undertaking study procedures
* History of current active malignancy as per investigator discretion other than breast cancer.
* Known or expected hypersensitivity to 68Ga NeoB

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — women with ER/PR+ HER2 - metastatic breast cancer
Enrollment: 20 (Estimated)
Dates: Start 2023-02-20 (Actual); Primary Completion 2025-02-20 (Estimated); Study Completion 2025-02-23 (Estimated)

PRIMARY OUTCOMES:
Assessment of Diagnostic Accuracy using a standard of truth (Biopsy, response to treatment RECIST and correlate images) | 2 years
  Diagnostic accuracy will be assessed by comparing lesions found on 68Ga NeoB PET CT to lesions found on conventional imaging (including CT, bone scan, and 18F-FDG PET/CT). Correlating images by sensitivity, specificity, true positive and negative predictive value

SECONDARY OUTCOMES:
Comparison of SUVmax/mean | 2 years
  To compare SUV max/mean of 68Ga- NeoB imaging to 18F-FDG PET CT in patients with metastatic ER/PR+ HER2- breast cancer.
Quantitative Variation in Lesion measuring total tumor volume and lesional intensity | 2 years
  By direct comparison of sites of known metastatic disease between 68Ga NeoB and conventional imaging. Assessing the presence and/or absence of lesions using SUVmax/SUVmean)
Comparison of variation in total tumour volume | 2 years
  To compare total tumour volume of 68Ga- NeoB imaging to 18F-FDG PET CT in patients with metastatic ER/PR+ HER2- breast cancer.

CONTACTS AND LOCATIONS:
Overall Officials: Louise Emmett, MD, Principal Investigator — St Vincent's Hospital, Sydney
Locations (1):
- St Vincent's Hospital, Sydney, New South Wales, Australia

IPD SHARING:
Plan to Share IPD: No
Results from both the 68NeoB PET CT and conventional imaging will be provided to the referring physician. It will be made clear to the physician that the 68NeoB PET results are experimental prior to participant enrolment. While the findings of the experimental agent are conveyed to the treating clinician, it is made clear that the results are experimental and should not be used for clinical purposes.